CLINICAL TRIAL: NCT06033157
Title: The Effect of Physiotherapist Supervised Training on Neuromuscular Control in Patients With Traumatic Anterior Shoulder Instability
Brief Title: Physiotherapist Supervised Training in Patients With Anterior Shoulder Instability
Acronym: ASIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristine Rask Andreasen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASIST-1
Record Dates: First submitted 2023-08-16; First posted 2023-09-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Shoulder Instability Subluxation Bilateral

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Active Comparator): A 12 week physiotherapist supervised training program
  Interventions: Behavioral: Physiotherapist supervised training
- No-training (No Intervention): A short consultation with a designated orthopedic surgeon and a folder with general advice on how to avoid further dislocations and to relieve pain from the shoulder.

INTERVENTIONS:
Behavioral: Physiotherapist supervised training — A 12 week physiotherapist supervised training program. The patient will receive supervision by a physiotherapist 6 times during the intervention period.
  The patient is strongly encouraged to do the assigned training protocol at home 3 times a week. The supervised physiotherapy consists of introduction, review and progression of the assigned exercises. In addition, the patient will receive education and guidance in daily use of the arm and appropriate load on the shoulder.
  Arms: Training

SUMMARY:
The goal of this clinical trial is to investigate if physiotherapist supervised training improves neuromuscular control in patients suffering from traumatic anterior shoulder instability. The main question(s) it aims to answer are:

* Does physiotherapist supervised training improve shoulder neuromuscular control
* Does physiotherapist supervised training prevent recurring shoulder dislocations
* Is physiotherapist supervised training as good as surgery in improving shoulder neuromuscular control Participants will be randomised to either a training group or a no-training group.

Participants in the training group will undergo a 12 week training-program supervised by a physiotherapist.

Participants in the no-training group will receive a consultation with a shoulder surgeon, where information and general advice regarding the shoulder injury is provided.

Researchers will compare the training group to the no-training group to see if physiotherapist supervised training improves shoulder neuromuscular control in patients with traumatic anterior shoulder instability. The training group will also be compared to a historic group of patients with traumatic anterior shoulder instability, who underwent arthroscopic surgery.

DETAILED DESCRIPTION:
* Aim: To investigate the effect of physiotherapist supervised training on shoulder neuromuscular control, and increase understanding of traumatic anterior shoulder instability.
* Main research questions:

A: Is supervised training in patients with traumatic anterior shoulder instability better in improving neuromuscular control, strength, apprehension and patient reported outcomes when compared to no training.

B: Is supervised training in patients with traumatic anterior shoulder instability better in preventing re-dislocations and need for surgical stabilisation when compared to no training.

C: Is supervised training in patients with traumatic anterior shoulder as good as Bankart surgery in improving neuromuscular control and patient reported outcome when compared to no training.

• Objectives for research question A:

To investigate if, in patients with traumatic anterior shoulder instability, a supervised 12-week training programme is better than no training in improving:

1. Neuromuscular control
2. Shoulder internal rotational strength
3. Shoulder apprehension
4. Patient reported outcomes
5. Clinical shoulder instability Outcomes are measured at a) the end of the 12-weeks intervention and b) 6 months after the beginning of the intervention. Furthermore, patient reported outcomes is also measured at 1 and 2 years after the beginning of the intervention.

   * Objective for research question B:

To investigate if, in traumatic anterior shoulder instability, a supervised 12-week training programme is better than no training in preventing a) re-dislocations and b) need for surgical stabilisation within the first 24 months.

• Objectives for research question C:

To investigate if, in patients with traumatic anterior shoulder instability, a specialised 12-week training programme is as good as arthroscopic Bankart surgery in improving:

1. Neuromuscular control
2. Shoulder internal rotational strength
3. Shoulder apprehension
4. Patient reported outcomes The training group is measured 6 months after the beginning of the intervention and the historic Bankart surgery group is measured 6 months after the surgery.

For all objectives neuromuscular control is investigated by determining a) shoulder joint position sense (JPS), b) shoulder reaction time, and c) shoulder sway length.

* Type of study: Pilot randomized controlled trial including 64 patients, which is allocated to either training og no-training (32 patients in each group).
* Time schedule: Recruitment and inclusion is planned to begin September 1st 2023 and is expected to last for 12-18 months. With a 2-year follow-up the complete study period is expected to last 3-3,5 years.
* Set-up: Patients presenting with shoulder instability in the outpatient clinic at Department of Orthopedic Surgery, Copenhagen University Hospital Hvidovre, will be recruited for the study. Patients who have signed an informed consent form will be randomised to either training- og no training-intervention and undergo examinations prior to, as well as three and six months after beginning of the intervention. All examinations will take place at the Copenhagen University Hospital Hvidovre. Patients in the training-group will be refered to training supervised by a physiotherapist. The training will take place at either Copenhagen University Hospital Hvidovre or a municipal rehabilitation center in Copenhagen. All examinations will include neuromuscular testing, accompanied by a clinical shoulder examination, strength measures and a validated electronic questionnaires regarding shoulder-related function. A pre-interventional 3D computed tomography scan will be performed to evaluate bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* Unilateral traumatic anterior shoulder instability.
* Willingness to adhere to the study protocol, herein attend follow-up.
* Ability to speak, read, and understand Danish.
* Ability to give written informed consent.

Exclusion Criteria:

* Instability in the opposite shoulder.
* Off-track lesion.
* For both shoulders: Former or planned surgery.
* For both shoulders: posterior, multi-directional or atraumatic instability.
* For both shoulders: traumatic rotator cuff or biceps tendon tear.
* For both shoulders: traumatic fracture of proximal humerus (other than Hill-Sachs lesion), clavicula, scapula (other than glenoid) or dislocation of sternoclavicular or acromioclavicular joints.
* For both shoulders: atraumatic shoulder pathologies (e.g. frozen shoulder, symptomatic osteoarthritis of the shoulder or acromioclavicular joints, acute tendinitis calcarean).
* Pregnancy.
* Terminal illness or severe medical illness: ASA score ≥3.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular control - Shouldersway | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  - Shoulder sway. Measured as sway-length (in millimeter).

SECONDARY OUTCOMES:
Clinical examination - Shoulder instability | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  - Shoulder instability tests: Sulcus sign, load and shift, apprehension test, relocation test.
Clinical examination - Shoulder range of motion | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  - Shoulder range of motion in flexion, extension, abduction, internal and external rotation
Strength measure | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  Shoulder internal rotational strength, measured in Newton.
Apprehension measure | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  An assessment (in degree) of when during an external rotational movement, the patient feels apprehension.
Patient-reported outcome measures | Will be tested prior to intervention and 3, 6, 12 and 24 months after the beginning of the intervention
  * WOSI-score
  * Purpose-made questions about return to sport and work, and fear of reinjury.
Redislocations | Will be tested 3, 6, 12 and 24 months after the beginning of the intervention
  Patients will be asked on every visit, if they have sustained re-dislocation of their shoulder
Neuromuscular control - Joint Position Sense | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  - Joint position sense for shoulder external rotation. Repositioning error is measured in degree.
Neuromuscular control - Reaction Time | Will be tested prior to intervention and 3 and 6 months after the beginning of the intervention
  - Reaction time. Measured as the time (in milliseconds) it takes the patient to respond to a sudden movement in the shoulder joint.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine R Andreasen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre; Kristoffer W Barfod, MD, PhD, Study Chair — Copenhagen University Hospital, Hvidovre; Kristoffer W Barfod, MD, PhD, Study Director — Copenhagen University Hospital, Hvidovre
Locations (1):
- Sports Orthopedic Research Center - Copenhagen (SORC-C), Department of Orthopedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No